CLINICAL TRIAL: NCT04248036
Title: Trygghetscirkelns föräldraskap (Circle of Security - Parenting) - Gruppintervention för föräldrar Med Barn förskoleåldern - En Pilotstudie.
Brief Title: Circle of Security - Parenting, COS-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VGFOUSA-903421
Record Dates: First submitted 2020-01-19; First posted 2020-01-30 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-09

CONDITIONS: Parenting; Psychological Phenomena and Processes; Primary Health Care
Keywords: Parenting

STUDY DESIGN:
Intervention Model Description: Pilot study
Masking Description: Group Care providers are masked for outcome assesment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Circle Of Security Parenting, COS-P (Other): Pilot study, assessing eligibility, outcome measures and compliance to Group intervention
  Interventions: Behavioral: Circle of Security - Parenting, COS-P

INTERVENTIONS:
Behavioral: Circle of Security - Parenting, COS-P — Circle of Security - Parenting is a manual-based, psychoeducational intervention program in group that includes 8 group sessions of 90 minutes each.

SUMMARY:
Background: Circle of Security-Parenting is a parental support program that provides basic knowledge about the emotional needs of children up to 6 years old and is illustrated graphically based on a circle model. It is designed to be given in group and includes 8 sessions of 90 minutes each.

COS-P is regularly offered as a parent support intervention within the Psychology units for Maternal and Child health care in Södra Älvsborg and Fyrbodal with the aim of increasing the quality of the parent-child relationship.

Objective: Prior to a planned RCT study, clarify which inclusion criterias are used for the COS-P intervention within the two psychology units, which parents accept and complete the study and investigate change in self-assessed depression, anxiety and stress level in the parent, the parent's reflective ability and symptoms in the child estimated by the parent.

Method: The parents who participate in the planned COS-P groups within the two units in spring/autumn of 2020 will fill in surveys before group start, at the end of intervention and 6-months follow up. Change between baseline and posttest as well as between baseline and 6-month follow-up will be analyzed.

The psychologists will fill in specially formulated questionnaires regarding their inclusion criterias.

Expected result: This pilot study is expected to describe the group of parents receiving COS-P and the inclusion criterias for the intervention used by the psychologists in the Psychology units for Maternal and Child health care in Södra Älvsborg and Fyrbodal.

DETAILED DESCRIPTION:
Background: Circle of Security-Parenting (COS-P) is a manual-based, psychoeducational parental support program that includes 8 group sessions of 90 minutes each. It provides basic knowledge about the emotional needs of children up to 6 years old and how parents can meet those needs to promote secure attachment in their child.

COS-P is a parental support groupintervention that is regularly given in the Psychology units for Maternal and Child health care in Södra Älvsborg and Fyrbodal and has become an appreciated intervention by both the participants and the psychologists who lead the groups. The method is also increasingly used both in Sweden and internationally but the systematic evaluation of COS-P is at the same time very limited. It is also unclear what the inclusion criterias and outcome measures are for COS-P in the Psychology unit for Maternal and Child health care.

Objective: The purpose of this pilot study is to provide knowledge of the inclusion criterias and outcome measures for COS-P within the Psychological units for Maternal and Child health care in Södra Älvsborg and Fyrbodal before more research subjects and activities are included in a randomized controlled study. The study also aims to examine change in the participating parents between baseline and posttest as well as the 6-month follow-up regarding self-assessed depression, anxiety and stress level, the parent's reflective ability and symptoms in the child estimated by the parent.

Additionally, the study will describe whether there is a relationship between demographic data and self-assessed depression, anxiety, stress level, the parent's reflective ability and symptoms of the child estimated by the parent at baseline and posttest and at baseline and 6-month follow-up.

Method: The parents who are assessed suitable for COS-P and accept to participate in the pilot study during spring/autumn 2020 will fill in surveys before group start, after completion and at the 6-month follow-up. In total, 50 parents will be included in the study.

Psychologists will fill in specially formulated questionnaires regarding their inclusion criterias.

Expected result: This pilot study is expected to describe the group of parents receiving COS-P and the inclusion criterias for the intervention used by the psychologists in the Psychology units for Maternal and Child health care in Södra Älvsborg and Fyrbodal.

ELIGIBILITY:
Inclusion criteria:

* The parent has difficulties in understanding and/or reflecting upon the childs signals/emotional needs.
* The parent has diffuculties in bonding to the child.
* The parent has difficulties in helping the child with emotional regulation.

Exclusion criteria:

* Serious mental illness
* Lack of language skills in Swedish.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Short term effect of COS-P on parental reflective functioning. | Change from baseline to completion of intervention, an average of 8-12 weeks.
  What is the effect of COS-P on the parent´s capacity to reflect upon both his/her own internal mental experiences and those of the child measured by change in scores in "The Parental Reflective Functioning Questionnaire", the 18 items version, from baseline to posttest?
Short term effect of parent´s participation in COS-P on the child´s behavioral problems/mental health. | Change from baseline to completion of intervention, an average of 8-12 weeks.
  What is the effect of the parent´s participation in COS-P on the child´s behavioral problems/mental health measured by change in scores in "The Strengths and Difficulties Questionnaire (SDQ) for preschool Children" from baseline to posttest..
Long term effect of COS-P on parental reflective functioning. | Change from baseline to 6-month follow-up.
  What is the effect of COS-P on the parent´s capacity to reflect upon both his/her own internal mental experiences and those of the child measured by change in scores in "The Parental Reflective Functioning Questionnaire", the 18 items version, from baseline to 6-month follow-up?
Long term effect of parent´s participation in COS-P on the child´s behavioral problems/mental health. | Change from baseline to 6-month follow-up.
  What is the effect of the parent´s participation in COS-P on the child´s behavioral problems/mental health measured by change in scores in "The Strengths and Difficulties Questionnaire (SDQ) for preschool Children" from baseline to 6-month follow-up?

SECONDARY OUTCOMES:
Short term effect of COS-P on parental stress level. | Change from baseline to completion of intervention, an average of 8-12 weeks.
  What is the effect of COS-P on parental stress level measured by change in scores in "Swedish Parenthood Stress Questionnaire" from baseline to posttest?
Short term effect of COS-P on depressive mood in parent. | Change from baseline to completion of intervention, an average of 8-12 weeks.
  What is the effect of COS-P on depressive mood in parent measured by change in scores in "Beck Depressive Inventory - 2" from baseline to posttest?
Short term effect of COS-P on anxiety in parent. | Change from baseline to completion of intervention, an average of 8-12 weeks.
  What is the effect of COS-P on anxiety in parent measured by change in scores in "Beck Anxiety Inventory" from baseline to posttest?
Long term effect of COS-P on parental stress level. | Change from baseline to 6-month follow-up.
  What is the effect of COS-P on parental stress level measured by change in scores in "Swedish Parenthood Stress Questionnaire"?
Long term effect of COS-P on depressive mood in parent. | Change from baseline to 6-month follow-up.
  What is the effect of COS-P on depressive mood in parent measured by change in scores in "Beck Depressive Inventory - 2" from baseline to 6-month follow-up?
Long term effect of COS-P on anxiety in parent. | Change from baseline to 6-month follow-up.
  What is the effect of COS-P on anxiety in parent measured by change in scores in "Beck Anxiety Inventory" from baseline to 6-month follow-up?

OTHER OUTCOMES:
A questionnaire designed for the psychologists in the study containing 4 specific questions. | Through study completion, an average of 1 year.
  1. "What inclusion criterias did you use when you offered a parent to participate in COS-P?"
  2. "How many parents have you offered the opportunity to participate in COS-P over the past 6 months?"
  3. "How many of these have accepted to participate in COS-P?"
  4. "What other intervention have you offered to those parents who have declined to participate in COS-P?"

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye Sag, BSc, Principal Investigator — Regionhälsan, Region Västra Götaland
Locations (1):
- Psykologenheten för mödra- och barnhälsovården, Gothenburg, Västra Götaland County, Sweden